CLINICAL TRIAL: NCT06069557
Title: The Effect of Respiratory Exercises and Incentive Spirometer Use in the Early Postoperative Period on Abdominal Distension, Shoulder Pain and Mobilization Process in Laparoscopic Cholecystectomy Patients
Brief Title: The Effect of Respiratory Exercises on Abdominal Distension in Laparoscopic Cholecystectomy Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Araz ASKEROĞLU, Assoc. Prof. Dr., Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21415022005
Record Dates: First submitted 2023-09-29; First posted 2023-10-06 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Elective Laparoscopic Cholecystectomy
Keywords: Laparoscopic cholecystectomy; Pneumoperitoneum; Shoulder pain; Deep breathing exercises; incentive spirometry
MeSH Terms: conditions — Pneumoperitoneum; Shoulder Pain | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: In our study, there are two groups, one control group and one experimental group. The control group will not be intervened. The experimental group will receive preoperative training about the postoperative intervention and the effect of the intervention will be evaluated in postoperative period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): There will be no intervention in this group.
- Experimental (Experimental): An intervention will be made to this group
  Interventions: Other: Respiratory exercise

INTERVENTIONS:
Other: Respiratory exercise — This group will undergo intervention. The participants will be assessed in terms of abdominal distension and shoulder pain in preoperative period. Respiratory exercise training will be given in the preoperative period. At the 1st, 2nd, 3rd, 4th, 5th, 4th, 5th, and 6th hours postoperatively, 10 deep breathing exercises will be performed in semi fowlers 45º position. During this 6-hour period, the patient will be asked to give 10 deep breaths into the incentive spirometer every 2 hours. Patients will be evaluated for abdominal distension and shoulder pain at the 1st, 2nd, 3rd, 4th, 5th, and 6th hours postoperatively and mobilization times will be measured in the first 6 hours.
  Arms: Experimental

SUMMARY:
Laparoscopic cholecystectomy is the first-line treatment for symptomatic gallstones. Pneumoperitoneum is the process of expanding the abdominal cavity during the surgical procedure by introducing CO2 gas into the abdomen to widen the field of view and operation. Although CO2 gas is usually released through the subumbilical incision at the end of laparoscopic cholecystectomy, some CO2 gas remains in the peritoneal cavity. This CO2 gas remaining in the peritoneal cavity can cause abdominal distension. Abdominal distension may also increase postoperative pain. In a study, abdominal distension was observed in 42.7% of patients who underwent laparoscopic surgery under general anesthesia. Although CO2 gas is usually released through the subumbilical incision at the end of laparoscopic cholecystectomy, some CO2 gas remains in the peritoneal cavity. This CO2 gas remaining in the peritoneal cavity may cause abdominal distension. On the other hand the incidence of shoulder pain due to pneumoperitoneum and CO2 insufflation after laparoscopic surgery ranges from 35% to 60%. In a study conducted in the Republic of Korea in 2016 in 105 laparoscopic surgery patients, the incidence of shoulder pain after laparoscopy was found to be 80% in the first 24 hours. Inappropriate treatment of postoperative pain in laparoscopic surgery can lead to delayed mobilization, patient dissatisfaction, delayed hospital discharge, and development of chronic pain. In this study, the effect of respiratory exercises and the use of incentive spirometry in the early postoperative period on abdominal distension, shoulder pain and mobilization process in laparoscopic cholecystectomy patients will be examined. We aimed to evaluate the effect of deep breathing exercises and the use of incentive spirometry in the early postoperative period on abdominal distension and shoulder pain due to insufflation procedure in laparoscopic cholecystectomy patients. It is important to take some precautions from the early period to prevent problems that may develop after abdominal surgery. It is thought that the use of deep breathing exercises and incentive spirometry in the early period after laparoscopic cholecystectomy will have an effect on abdominal distension, shoulder pain and mobilization process due to the insufflation procedure.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is the removal of the cystic duct or dissection of the gallbladder with the help of 4 trocar incision lines and intraoperative cholangiography by creating pneumoperitoneum with Veress needle or Hasson technique while the patients are under general anesthesia. Pneumoperitoneum is the process of expanding the abdominal cavity during the surgical procedure by introducing CO2 gas into the abdomen to widen the field of view and operation. With high-pressure insufflators, CO2 is introduced into the abdomen at an intra-abdominal pressure of 15mmHg. The increase in abdominal pressure caused by abdominal distension affects circulation and ventilation by acting directly on the abdominal compartment and indirectly on the thoracic compartment. The increase in abdominal pressure caused by abdominal distension affects circulation and ventilation by acting directly on the abdominal compartment and indirectly on the thoracic compartment. In a study, abdominal distension was observed in 42.7% of patients who underwent laparoscopic surgery under general anesthesia. Although CO2 gas is usually released through the subumbilical incision at the end of laparoscopic cholecystectomy, some CO2 gas remains in the peritoneal cavity. This CO2 gas remaining in the peritoneal cavity may cause abdominal distension. Abdominal distension may also increase postoperative pain. A study results showed that patients with high abdominal distension had higher average postoperative pain levels during the recovery period. It was also found that patients with high levels of postoperative pain caused a delay in readiness for discharge from the recovery room. In addition, inappropriate treatment of postoperative pain in laparoscopic surgery can lead to delayed mobilization, patient dissatisfaction, delayed hospital discharge, and development of chronic pain. Pulmonary atelectasis, decrease in functional residual capacity and high peak airway pressures may occur due to CO2 ensufflation. In addition, an increase in central venous pressure and an increase in arterial and alveolar CO2 can be detected due to increased intra-abdominal pressure and CO2 absorption. Pulmonary complication rates may reach 20% after upper abdominal and thoracic operations, especially due to decreased use of the diaphragm because of pain. In the literature, it was seen that the most common intervention applied after surgery as a nursing practice in the elimination of abdominal distension was to stand up the patient and to make active and passive movements in the bed. Early mobilization, frequent position changes, deep breathing and coughing exercises, and hydration are important in preventing complications that may develop in the respiratory system. The aim of deep breathing exercises is to ensure deep breathing after surgery and to obtain normal breathing patterns.The incentive spirometer is used to assess the patient's inspiratory effort by measuring the volume of inhalation. The incentive spirometer can be used as a convenient tool in rehabilitation as it is inexpensive and easy to administer with no known side effects. It is thought that the use of deep breathing exercises and incentive spirometry in the early period after laparoscopic cholecystectomy will have an effect on abdominal distension, shoulder pain and mobilization process due to the insufflation procedure.

ELIGIBILITY:
Inclusion Criteria:

Volunteer Aged between 18-65 years Comprehensible verbal communication

Exclusion Criteria:

Patients with hearing problems Unstable hemodynamics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 18-65
Enrollment: 156 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Post operative abdominal distension | Postoperative 1st, 2nd, 3rd, 4th, 4th, 5th, and 6th hours.
  In the postoperative period, after the patients come to the clinic, all patients will be examined for abdominal distension and their abdominal circumferences will be measured with a tape measure and will be compared with the preoperative period. Patient's statement will also be asked.

SECONDARY OUTCOMES:
Post operative shoulder pain | Postoperative 1st, 2nd, 3rd, 4th, 4th, 5th, and 6th hours.
  In the postoperative period, all patients' shoulder pain will be measured with with the Numeric Pain Rating Scale (NPRS) after the patients come to the clinic. The scale is typically set up on a horizontal line, ranges most commonly from 0-10. Patients are instructed to choose a single number from the scale that best indicates their level of pain.
Mobilization time | The first 6 hours in the early postoperative period.
  Mobilization times will be measured in minutes in the first 6 hours in the early postoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Araz Askeroğlu, Ph.D., Principal Investigator — Çanakkale Onsekiz Mart University
Locations (1):
- Bursa City Hospital, Bursa, Bursa Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aydemir O, Aslan FE, Karabacak U, Akdas O. Corrigendum to 'The Effect of Exaggerated Lithotomy Position on Shoulder Pain after Laparoscopic Cholecystectomy' Pain Management Nursing 2018;19(6):663-670. Pain Manag Nurs. 2019 Feb;20(1):89. doi: 10.1016/j.pmn.2019.01.002. No abstract available. PMID 30782392
- [Result] Bataineh AM, Qudaisat IY, Banihani M, Obeidat R, Hamasha HS. Use of intraoperative mild hyperventilation to decrease the incidence of postoperative shoulder pain after laparoscopic gastric sleeve surgery: A prospective randomised controlled study. Indian J Anaesth. 2021 Nov;65(11):806-812. doi: 10.4103/ija.ija_576_21. Epub 2021 Nov 23. PMID 35001953
- [Result] Alaparthi GK, Augustine AJ, Anand R, Mahale A. Comparison of Diaphragmatic Breathing Exercise, Volume and Flow Incentive Spirometry, on Diaphragm Excursion and Pulmonary Function in Patients Undergoing Laparoscopic Surgery: A Randomized Controlled Trial. Minim Invasive Surg. 2016;2016:1967532. doi: 10.1155/2016/1967532. Epub 2016 Jul 21. PMID 27525116
- [Result] Hsu KF, Chen CJ, Yu JC, Wu SY, Chen BC, Yang CW, Chen TW, Hsieh CB, Chan DC. A Novel Strategy of Laparoscopic Insufflation Rate Improving Shoulder Pain: Prospective Randomized Study. J Gastrointest Surg. 2019 Oct;23(10):2049-2053. doi: 10.1007/s11605-018-3896-5. Epub 2018 Oct 8. PMID 30298416
- [Result] Tuvayanon W, Silchai P, Sirivatanauksorn Y, Visavajarn P, Pungdok J, Tonklai S, Akaraviputh T. Randomized controlled trial comparing the effects of usual gas release, active aspiration, and passive-valve release on abdominal distension in patients who have undergone laparoscopic cholecystectomy. Asian J Endosc Surg. 2018 Aug;11(3):212-219. doi: 10.1111/ases.12451. Epub 2017 Dec 20. PMID 29266752
- [Result] Yi MS, Kim WJ, Kim MK, Kang H, Park YH, Jung YH, Lee SE, Shin HY. Effect of ultrasound-guided phrenic nerve block on shoulder pain after laparoscopic cholecystectomy-a prospective, randomized controlled trial. Surg Endosc. 2017 Sep;31(9):3637-3645. doi: 10.1007/s00464-016-5398-4. Epub 2016 Dec 30. PMID 28039653
- [Result] Zeeni C, Chamsy D, Khalil A, Abu Musa A, Al Hassanieh M, Shebbo F, Nassif J. Effect of postoperative Trendelenburg position on shoulder pain after gynecological laparoscopic procedures: a randomized clinical trial. BMC Anesthesiol. 2020 Jan 29;20(1):27. doi: 10.1186/s12871-020-0946-9. PMID 31996139